CLINICAL TRIAL: NCT00371241
Title: Antibody Secreting Cell (ASC) and Immunoactive Protein Profiles in Neonates on Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Antibody Secreting Cell and Cyotokine Profiles in Neonates on ECMO
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Hospital (Other)
Responsible Party: James R. Murphy, The University of Texas Health Science Center, HoustonU
Other Study IDs: HSC-MS-06-0122
Record Dates: First submitted 2006-08-30; First posted 2006-09-04 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Persistent Fetal Circulation Syndrome; Diaphragmatic Hernia; Meconium Aspiration; Sepsis
Keywords: ECMO; extracorporeal membrane oxygenation; cytokines; chemokines
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome; Hernia, Diaphragmatic; Meconium Aspiration Syndrome; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Infants are placed on ECMO for correction of reversible respiratory failure. Often, because a few of the reasons for respiratory failure show us similar things in the baby, it is difficult to determine exactly which is causing the biggest problem. We are now capable of measuring certain cells and proteins in these infants that may help us more accurately diagnose the exact problem. We hypothesize that infants placed on ECMO will show unique antibody-secreting cells responses and patterns of cytokine and chemokine (protein) response to illness and to the ECMO circuit. If we find unique patterns to these cells or proteins, they may be able to predict outcomes or guide treatment of these infants.

DETAILED DESCRIPTION:
Specific Aims Primary Objective

1. Determine the rise, peak, and fall of immunoglobulin isotype-specific ASC's, and immunoactive proteins (cytokines and chemokines) from sequential samples of peripheral blood from infants on ECMO.

Secondary Objectives:

1. Determine the most appropriate time to sample blood from infants with suspected sepsis for ASC diagnostic assay.
2. Characterize the incidence of culture-negative sepsis that leads to ECMO.
3. Determine immunoglobulin isotype-specific levels of ASC in infants with and without infection.
4. Establish an archive of mononuclear cells and plasma to use in development of pathogen specific ASC assays.

Hypothesis Infants on ECMO will have a high ASC response and unique cytokine/chemokine patterns due to possible underlying infection and exposure to many foreign antigens (blood products, ECMO circuit). A significant portion of these will have ASC's with specificity for common causes of neonatal sepsis that is not detected by routine blood culture.

Procedures:

Residual samples will be collected from those used in routine procedures for infants on ECMO. The approximate volume/sample will be 0.5-0.8ml. Specimens will be processed using methods well established in our laboratory. Briefly, PBMC's will be isolated via Ficoll gradient and archived in liquid nitrogen at -80C. Batch analysis of ASC levels and lymphocyte proliferation activity will be performed when sufficient number of specimens are accumulated. A detailed profile and quantification of immune cells will be determined by Fluorescent Activated Cell Sorter (FACS) staining for CD3, CD4, CD8, CD27, CD38, CD45, and HLA-DR. A bead micro-array will be used to detect levels of immunoactive molecules, also done on the FACS. The proteins detected will include, but may not be limited to, the following: IL1β, IL2, IL4, IL5, IL6, IL7, IL8, IL10, IL12p70, IL13, IL17, GCSF, GMCSF, IFN-γ, MCP-1, MIP-1β, TNFα. The ASC procedure be that established by Van de Verg modified to use membrane surface microculture plates in place of agar with outcomes read by CTL analyzer in place of manual count. LPA assays will use long established techniques.

ELIGIBILITY:
Inclusion Criteria:

* 1) term newborn infants >24 hours and ≤ 30 days old 2) Placed on ECMO in the NICU at MHCH 3) Parental consent obtained within 48 hours of being placed on ECMO

Exclusion Criteria:

* 1) Infant > 30 days old 2) Infant NOT on ECMO 3) Withdrawal of parental consent

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants requiring ECMO
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2006-09; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Murpy, PhD, Principal Investigator — University of Texas Health Science Center at Houston- Division of Infectious Diseases
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Stoll BJ, Lee FK, Hale E, Schwartz D, Holmes R, Ashby R, Czerkinsky C, Nahmias AJ. Immunoglobulin secretion by the normal and the infected newborn infant. J Pediatr. 1993 May;122(5 Pt 1):780-6. doi: 10.1016/s0022-3476(06)80026-0. PMID 8496761
- [Background] Stoll BJ, Lee FK, Larsen S, Hale E, Schwartz D, Rice RJ, Ashby R, Holmes R, Nahmias AJ. Clinical and serologic evaluation of neonates for congenital syphilis: a continuing diagnostic dilemma. J Infect Dis. 1993 May;167(5):1093-9. doi: 10.1093/infdis/167.5.1093. PMID 8486942
- [Background] Baqar S, Nour El Din AA, Scott DA, Bourgeois AL, Mourad AS, Kleinosky MT, Oplinger MJ, Murphy JR. Standardization of measurement of immunoglobulin-secreting cells in human peripheral circulation. Clin Diagn Lab Immunol. 1997 May;4(3):375-9. doi: 10.1128/cdli.4.3.375-379.1997. PMID 9144380
- [Background] Kuster H, Weiss M, Willeitner AE, Detlefsen S, Jeremias I, Zbojan J, Geiger R, Lipowsky G, Simbruner G. Interleukin-1 receptor antagonist and interleukin-6 for early diagnosis of neonatal sepsis 2 days before clinical manifestation. Lancet. 1998 Oct 17;352(9136):1271-7. doi: 10.1016/S0140-6736(98)08148-3. PMID 9788457